CLINICAL TRIAL: NCT00341770
Title: Assessment of Sympathetic Nervous System Activity by Microneurography Recording Technique
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999910107; OH91-DK-0107
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-23

CONDITIONS: Nervous System
MeSH Terms: conditions — Neurologic Manifestations

SUMMARY:
Obesity is the consequence of an imbalance between energy intake and energy expenditure. Recent studies have suggested that the sympathetic nervous system (SNS) may be an important determinant of the rate of energy expenditure in man. Indirect assessments of the sympathetic nervous activity in Pima Indians have recently shown impaired SNS-mediated energy expenditure in this obesity-prone population. We plan to perform direct microelectrode nerve recording of the sympathetic innervation of the lower leg to directly assess SNS activity and examine its potential role in the regulation of metabolic rate and the development of obesity. Measurements will be performed in the basal state, in response to glucose feeding (75 g OGTT) and in response to glucose/insulin infusion. These studies also will help to disassociate the effect of insulin and glucose on the stimulation of SNS activity. Energy expenditure measurements will be performed over 24 hours in the respiratory chamber and for 2 1/2 hours before and during the euglycemic clamp. Results also will be used to determine possible racial differences between Pimas and Caucasians, since the risk for obesity is markedly different in these populations. To exclude the possibility of a "normal" SNS activity but with peripheral resistance to the action of norepineprine, we will perform adrenergic stimulation by isoproterenol to measure peripheral adrenergic sensitivity.

DETAILED DESCRIPTION:
Obesity is the consequence of an imbalance between energy intake and energy expenditure. Recent studies have suggested that the sympathetic nervous system (SNS) may be an important determinant of the rate of energy expenditure in man. Indirect assessments of the sympathetic nervous activity in Pima Indians have recently shown impaired SNS-mediated energy expenditure in this obesity-prone population. We plan to perform direct microelectrode nerve recording of the sympathetic innervation of the lower leg to directly assess SNS activity and examine its potential role in the regulation of metabolic rate and the development of obesity. Measurements will be performed in the basal state, in response to glucose feeding (75 g OGTT), in response to a standard meal, and in response to glucose/insulin infusion. These studies also will help to disassociate the effect of insulin and glucose on the stimulation of SNS activity. The association between postprandial changes in SNS activity and subjective ratings of hunger and fullness also will be studied. Energy expenditure measurements will be performed over 24 hours in the respiratory chamber and for 2 1/2 hours before and during the euglycemic clamp. Results also will be used to determine possible racial differences between Pimas and Caucasians, since the risk for obesity is markedly different in these populations. To exclude the possibility of a "normal" SNS activity but with peripheral resistance to the action of norepineprine, we will perform adrenergic stimulation by isoproterenol to measure peripheral adrenergic sensitivity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male and female Pima Indians, age 4 years old and older.

Male and female Caucasians, age 4 years old and older.

Offspring of Diabetic and Non-Diabetic mothers will be recruited.

Male and female monozygotic and dizygotic twins of any racial background between the ages of 4-7 will be considered for study.

Indian subjects will be recruited from the Gila River Indian Community.

Only children found in good health on the basis of the medical history and physical examination will be accepted into the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 1991-04-12; Study Completion 2010-11-23

CONTACTS AND LOCATIONS:
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Bray GA, York DA, Fisler JS. Experimental obesity: a homeostatic failure due to defective nutrient stimulation of the sympathetic nervous system. Vitam Horm. 1989;45:1-125. doi: 10.1016/s0083-6729(08)60393-3. PMID 2688303
- [Background] Ravussin E, Lillioja S, Knowler WC, Christin L, Freymond D, Abbott WG, Boyce V, Howard BV, Bogardus C. Reduced rate of energy expenditure as a risk factor for body-weight gain. N Engl J Med. 1988 Feb 25;318(8):467-72. doi: 10.1056/NEJM198802253180802. PMID 3340128
- [Background] O'Dea K, Esler M, Leonard P, Stockigt JR, Nestel P. Noradrenaline turnover during under- and over-eating in normal weight subjects. Metabolism. 1982 Sep;31(9):896-9. doi: 10.1016/0026-0495(82)90178-0. PMID 7121260